CLINICAL TRIAL: NCT00987649
Title: Evaluation of CA125 and HE4 Assays to Estimate the Risk of Ovarian Cancer in Patients Presenting to a General Surgeon or Obstetrician/Gynecologist With an Adnexal Mass
Brief Title: Ovarian Cancer Risk Estimation in Patients With Pelvic Mass
Status: Completed | Type: Observational
Sponsor: Fujirebio Diagnostics, Inc. (Industry)
Collaborators: Advanced Clinical Research Services, LLC (Other); ReSearch Pharmaceutical Services, Inc. (Industry)
Responsible Party: Rebecca Simamora, Director Clinical Affairs, Fujirebio Diagnostics, Inc.
Other Study IDs: FDI-15
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2011-02-09 (Estimated); Status verified 2011-02

CONDITIONS: Adnexal Mass; Ovarian Cancer
Keywords: pelvic mass; ovarian cancer; adnexal mass; CA125; HE4
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, Plasma, Urine
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether the Risk of Ovarian Cancer Algorithm (ROMA) is effective in the determination of a woman's risk of cancer when she is scheduled to have surgery to remove a pelvic mass.

After Informed Consent is obtained, an Initial Cancer Risk Assessment will be made. A blood sample will be collected within 30 days of the surgical procedure. Results of the surgical procedure will be collected and analyzed against the CA125 and HE4 results used in the calculation of the ROMA.

ELIGIBILITY:
Inclusion Criteria:

* Female, age ≥ 18 years
* Adnexal mass present documented by imaging
* Scheduled to undergo surgery based on a finding of adnexal mass (defined as a simple, complex or a solid ovarian cyst/or any mass in pelvis)
* Able to understand and willing to provide Informed Consent

Exclusion Criteria:

* Previous history of ovarian cancer
* Previous history of bilateral oophorectomy
* Currently known to be pregnant
* Unable to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is anticipated that approximately 10 general or specialty centers geographically dispersed throughout the United States will be utilized.
Sampling Method: Probability Sample
Enrollment: 512 (Actual)
Dates: Start 2009-10; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
1. A statistically higher number of cancer patients are correctly assigned by the combination of Initial Cancer Risk assessment and positive ROMA test result than by Initial Cancer Risk assessment alone | Blood draw within 30 days of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Richard Moore, MD, FACOG, FACS, Principal Investigator — Women & Infants Hospital Rhode Island
Locations (13):
- United States (13):
  - Scripps Clinic Carmel Valley, San Diego, California
  - Women's Clinic of Northern Colorado, Fort Collins, Colorado
  - OB/GYN Specialists of the Palm Beaches, Jupiter, Florida
  - University of South Florida Medical Center, Tampa, Florida
  - Woman's Hospital, Baton Rouge, Louisiana
  - Weill Medical College of Cornell University, New York, New York
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Women & Infants Hospital Rhode Island, Providence, Rhode Island
  - Chattanooga GYN-ONCOLOGY, Chattanooga, Tennessee
  - Jackson Clinic, Jackson, Tennessee
  - Adams Patterson Gynecology & Obstetrics, Memphis, Tennessee

REFERENCES:
- [Derived] Moore RG, Hawkins DM, Miller MC, Landrum LM, Gajewski W, Ball JJ, Allard WJ, Skates SJ. Combining clinical assessment and the Risk of Ovarian Malignancy Algorithm for the prediction of ovarian cancer. Gynecol Oncol. 2014 Dec;135(3):547-51. doi: 10.1016/j.ygyno.2014.10.017. Epub 2014 Oct 23. PMID 25449569
- See also: Information related to Fujirebio Diagnostics, Inc. — http://www.fdi.com